CLINICAL TRIAL: NCT03469804
Title: Essai de Phase II Multicentrique évaluant le Pembrolizumab Dans le Traitement de la Maladie de Kaposi Classique ou endémique
Brief Title: Phase II Multicentric Study of Pembrolizumab in Classic or Endemic Kaposi's Sarcoma
Acronym: KAPKEY
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P160601; 2016-003714-27 (EudraCT Number)
Record Dates: First submitted 2018-03-12; First posted 2018-03-19 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Kaposi Sarcoma; Progression, Disease
MeSH Terms: conditions — Sarcoma, Kaposi; Disease Progression | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: 2-stage phase II Simon's Optimal Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab (Experimental): Pembrolizumab Route: intravenous infusion Dose regimen: 200 mg per infusion every 3 weeks Duration of treatment: 6 months (8 cycles)
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Route: intravenous infusion Dose regimen: 200 mg per infusion every 3 weeks Duration of treatment: 6 months (8 cycles)

SUMMARY:
Classic and endemic Kaposi's sarcoma (KS) are lymphangio-proliferations associated with human herpes virus 8 (HHV8), which treatment is poorly codified. Chemotherapies give at best 30-60% of transient responses. While interferon responses are frequent, this drug is often poorly tolerated in elderly patients. Therefore new therapies are needed. Classic KS represents an ideal model for evaluating new drugs since patients do not receive concomitant immunosuppressive regimens nor antiviral therapies.

Pembrolizumab, an anti-PD1 monoclonal antibody has recently been shown to improve survival in several solid tumors. In KS few data are available on the role of PD1-PD-L1 axis. A significant PD-L1 expression on HHV8-associated pleural effusion lymphomas and on KS samples have been recently reported. Our experience in classical and endemic KS supports the role of this pathway with expression of PD-L1 by subpopulations of T cells but also NK cells in peripheral blood cells from these patients and expression of PD-L1 by tumor cells in KS lesions.

In this study we will evaluate the benefit and safety profile of pembrolizumab in classic and endemic KS.

ELIGIBILITY:
Inclusion Criteria:

* Classic or endemic histologically confirmed KS
* Progressive disease
* KS with more than 10 lesions or involving more than one limb segment or with involvement >3% body surface
* KS with at least 4 lesions ≥5mm
* KS with at least 1 other cutaneous tumor available for repeated pharmacodynamics evaluation and be willing to provide tissue from cutaneous biopsy of a tumor lesion
* At least 4 weeks washout for all KS specific therapies including chemotherapy and immunotherapy
* Provide written, informed consent prior to the performance of any study specific procedures
* Be ≥ 18 years of age on day of signing informed consent.
* Have a performance status of 0 or 1 on the ECOG Performance Scale.
* Demonstrate adequate organ function:

Hematological : Absolute neutrophil count (ANC) ≥1,000/mm3, Platelets ≥100,000 / mm3, Hemoglobin ≥ 9 g/dL Renal: Calculated creatinine clearance ≥40 mL/min (using Modification of diet in renal disease (MDRD) formula) Hepatic: AST (SGOT) and ALT (SGPT) ≤ 2.5xULN, serum total bilirubin ≤ 1.5xULN OR direct bilirubin ≤ ULN for subjects with total bilirubin levels >1.5xULN.

* Female subject of childbearing potential should have a negative serum pregnancy within 72 hours prior to receiving the first dose of study medication
* Have a health insurance

Exclusion Criteria:

* Has a known history of organ transplantation or HIV (HIV 1/2 antibodies detected at selection) Is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has KS with symptomatic visceral involvement unless no other therapeutic option is available Previously received treatments with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA4 antibody or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways.
* Has a known history of active infectious hepatitis, type B (HBsAg detected) or C (HCV RNA detected) or active TB (Tuberculosis Bacillus).
* Has an active infection requiring systemic therapy.
* Has hypersensitivity to pembrolizumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within last 4 weeks or who has not recovered (i.e., > Grade 1 at selection) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 3 weeks prior to study Day 1 or who has not recovered (i.e., > Grade 1 at selection) from adverse events due to a previously administered agent (Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study). (Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy).
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Patients with vitiligo, type I diabetes mellitus, hypothyroidism, psoriasis non requiring systemic treatment are permitted to enroll.
* Has active non-infectious pneumonitis or known history of non-infectious pneumonitis that required steroids, severe pulmonary disease or hypoxia
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, or not willing to use adequate contraceptive methods from study Visit 1 throughout the study period up to 120 days after the last dose of study therapy.
* Has received a live vaccine within 30 days prior to the first dose of trial treatment or while participating in the trial.
* Is currently participating or has participated in a study of an investigational agent within 4 weeks of the first dose of treatment.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Patient under guardianship or curators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-03-20 (Estimated); Study Completion 2020-09-20 (Estimated)

PRIMARY OUTCOMES:
Best Overall Response Rate (BORR) | 6 months
  Best Overall Response Rate (BORR) defined by the occurrence of complete response or partial response following AIDS Clinical Trials Group (ACTG) criteria recorded from the start of treatment until 6 months or the beginning of any other specific systemic therapy for KS if it occurs before 6 months

SECONDARY OUTCOMES:
Best overall response rate according to Physical Global Assessment (PGA) | 6 months
  Best overall response rate according to Physical Global Assessment (PGA) score until 6 months or the beginning of any other specific systemic therapy for KS if it occurs before 6 months
Response rate according to ACTG and PGA criteria | 3 months
Response rate according to ACTG and PGA criteria | 6 months
Response rate on number of lesions | 3 months
  Response rate on number of lesions and at best response as defined following ACTG criteria
Response rate on number of lesions | 6 months
  Response rate on number of lesions and at best response as defined following ACTG criteria
Response rate on the size of target lesions | 3 months
  Response rate on the size of target lesions and at best response as defined following ACTG criteria
Response rate on the size of target lesions | 6 months
  Response rate on the size of target lesions and at best response as defined following ACTG criteria
Response rate on tumor infiltration of target lesions | 3 months
  Response rate on tumor infiltration of target lesions and at best response as defined following ACTG criteria
Response rate on tumor infiltration of target lesions | 6 months
  Response rate on tumor infiltration of target lesions and at best response as defined following ACTG criteria
Response rate on lymphedema | 3 months
  Response rate on lymphedema (circumference, scale of 0 (absence) to 3 (painful or oozing)) at Month 3, Month 6 and at best response as defined following ACTG criteria
Response rate on lymphedema | 6 months
  Response rate on lymphedema (circumference, scale of 0 (absence) to 3 (painful or oozing)) at Month 3, Month 6 and at best response as defined following ACTG criteria
Time to response | 6 months
  Time to response defined as the time to first response recorded from the start of treatment
Time to progression | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Saint-Louis Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Delyon J, Biard L, Renaud M, Resche-Rigon M, Le Goff J, Dalle S, Heidelberger V, Da Meda L, Toullec L, Carcelain G, Mourah S, Caillat-Zucman S, Allain V, Battistella M, Lebbe C. PD-1 blockade with pembrolizumab in classic or endemic Kaposi's sarcoma: a multicentre, single-arm, phase 2 study. Lancet Oncol. 2022 Apr;23(4):491-500. doi: 10.1016/S1470-2045(22)00097-3. Epub 2022 Mar 10. PMID 35279271